CLINICAL TRIAL: NCT02577523
Title: A Multicenter, Parallel-group, Rater-blinded, Randomized Clinical Study Investigating the Efficacy, Safety, Tolerability and Pharmacokinetics of 2 Dosing Regimens of ND0612H [ ] in Subjects With Advanced Parkinson's Disease
Brief Title: A Clinical Study of Efficacy, Safety, Tolerability and PK of ND0612H in Subjects With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND0612H-006
Record Dates: First submitted 2015-10-06; First posted 2015-10-16 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ND0612 (Levodopa/Carbidopa solution) Dosing Regimen 1 (Experimental): Dosing Regimen 1 of ND0612 (Levodopa/Carbidopa solution) continuous SC infusion over 24 hours.
  Interventions: Drug: ND0612 (Levodopa/Carbidopa solution)
- ND0612 (Levodopa/Carbidopa solution) Dosing Regimen 2 (Experimental): Dosing Regimen 2 of ND0612 (Levodopa/Carbidopa solution) continuous SC infusion over 14 hours. Infusion started at wake-up time supplemented with an oral IR LD/CD tablet.
  Interventions: Drug: ND0612 (Levodopa/Carbidopa solution) + morning oral IR-LD/CD

INTERVENTIONS:
Drug: ND0612 (Levodopa/Carbidopa solution) — The total daily dose of levodopa/carbidopa 720/90 mg. Device: CRONO TWIN pump system.
  Other Names: Regimen 1 - 24-hr infusion
  Arms: ND0612 (Levodopa/Carbidopa solution) Dosing Regimen 1
Drug: ND0612 (Levodopa/Carbidopa solution) + morning oral IR-LD/CD — The total daily dose levodopa/carbidopa from ND0612 538/67 mg. Morning dose of oral IR-LD/CD 150/15 mg. Device: CRONO TWIN pump system.
  Other Names: Regimen 2 - 14-hr infusion
  Arms: ND0612 (Levodopa/Carbidopa solution) Dosing Regimen 2

SUMMARY:
This is a multicenter, parallel-group, rater-blinded, randomized clinical study in subjects with advanced PD investigating the efficacy, PK, safety and tolerability of continuous SC infusion of 2 dosing regimens of ND0612H, a solution of LD/CD delivered via a pump system as a continuous SC infusion, compared to standard oral LD/CD. After screening, subjects will undergo 1 day of standard oral LD/CD inpatient dosing followed by 2 days of inpatient treatment with 1 of 2 randomly allocated (1:1 randomization ratio) dosing regimens of ND0612H continuous SC infusion. Subjects will then continue on a maintenance dose of the assigned ND0612H dosing regimen for the next 25 days. A safety visit will be performed 4 weeks after the last SC administration of the study drug for a total of about 2.5 months of participation for each subject enrolled into the trial.

DETAILED DESCRIPTION:
This phase IIa randomized, controlled, parallel-group study will be conducted in 36 subjects with advanced PD who are treated with oral LD/CD at a stable dose and have predictable morning "OFF" periods and at least 2.5 hrs of daily "OFF" periods. The study will investigate the efficacy, PK, safety and tolerability of continuous SC infusion of 2 dosing regimens of ND0612H. Regimen 1 will employ continuous infusion for 24 hrs using a low infusion rate at night and a higher rate at daytime with supplemental administration of oral immediate release (IR) LD/CD in the mornings. During the inpatient period of about 3 days, the site staff will manage the administration and replacement of the infusions. On Day 4 subjects will be discharged home after they and their study partners have received training on the administration of the infusion. Subjects will then continue on a maintenance dose of the assigned ND0612 dosing regimen for the next 25 days. A safety visit will be performed 4 weeks after the last SC administration of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female PD subjects of any race aged 30 to 80 years who sign an Institutional Review Board/Ethics Committee (IRB/EC)-approved informed consent form (ICF).
2. PD diagnosis consistent with the UK Brain Bank Criteria.
3. Modified Hoehn & Yahr scale in "ON" state of stage ≤3.
4. Taking at least 4 doses/day of LD (or at least 3 doses/day of Rytary) and taking, or have attempted to take, at least 2 other classes of anti-PD medications in a therapeutic dose for at least 30 consecutive days each.
5. Subjects must be stable on their anti-PD medications for at least 30 days before Day 1.
6. Subjects may have had prior exposure to SC apomorphine injections/infusion but must have stopped administration at least 4 weeks before the screening visit. Treatment with apomorphine is prohibited during the entire ND0612H treatment period.
7. Must have a minimum of 2.5 hrs of "OFF" time per day with predictable early morning "OFF" periods as estimated by the subject.
8. Must have predictable and well defined early morning "OFF" periods with a good response to LD for treatment of the early morning "OFF" in the judgement of the investigator.
9. Mini Mental State Examination (MMSE) score >26.
10. No clinically significant medical, psychiatric or laboratory abnormalities which the investigator judges would be unsafe or non-compliant in the study.
11. Female subjects must be surgically sterile, postmenopausal (defined as cessation of menses for at least 1 year), or willing to practice a highly effective method of contraception. All female participants must be non-lactating and non-pregnant and have a negative urine pregnancy test at Screening and at Baseline. Female subjects of childbearing potential must practice a highly effective method of contraception (e.g., oral contraceptives, a barrier method of birth control [e.g., condoms with contraceptive foams, diaphragms with contraceptive jelly], intrauterine devices, partner with vasectomy), 1 month before enrollment, for the duration of the study, and 3 months after the last dose of study drug.
12. Willingness and ability to comply with study requirements

Exclusion Criteria:

1. Atypical or secondary parkinsonism.
2. Acute psychosis or hallucinations in past 6 months.
3. Any relevant medical, surgical, or psychiatric condition, laboratory value, or concomitant medication which, in the opinion of the Investigator or the eligibility reviewer, makes the subject unsuitable for study entry or potentially unable to complete all aspects of the study.
4. Prior neurosurgical procedure for PD, or duodopa treatment.
5. Subjects with a history of drug abuse or alcoholism within the past 12 months.
6. Clinically significant ECG rhythm abnormalities.
7. Renal or liver dysfunction that may alter drug metabolism including: serum creatinine >1.3 mg/dL, serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 x upper limit of normal (ULN), total serum bilirubin >2.5 mg/dL.
8. Subjects who are not willing to operate the pump system.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Salin, MD, Study Director — NeuroDerm Ltd.
Locations (11):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - QUEST Research Institute, Farmington Hills, Michigan
  - University of Cincinnati, Cincinnati, Ohio
- Medical University Innsbruck, Innsbruck, Austria
- Israel (3):
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (4):
  - University Foundation, Chieti
  - AOU Pisa, Pisa
  - IRCCS San Raffaele Pisana, Rome
  - Fondazione Ospedale San Camillo - I.R.C.C.S., Venice

REFERENCES:
- [Result] Olanow CW, Espay AJ, Stocchi F, Ellenbogen AL, Leinonen M, Adar L, Case RJ, Orenbach SF, Yardeni T, Oren S, Poewe W; 006 study group. Continuous Subcutaneous Levodopa Delivery for Parkinson's Disease: A Randomized Study. J Parkinsons Dis. 2021;11(1):177-186. doi: 10.3233/JPD-202285. PMID 33164945

RESULTS

PARTICIPANT FLOW:
Groups:
- ND0612 (Levodopa/Carbidopa Solution) Dosing Regimen 1: Dosing Regimen 1 of ND0612 (Levodopa/Carbidopa solution) continuous SC infusion over 24 hours
  ND0612 (Levodopa/Carbidopa solution, 720/90 mg daily)
- ND0612 (Levodopa/Carbidopa Solution) Dosing Regimen 2: Dosing Regimen 2 of ND0612 (Levodopa/Carbidopa solution) continuous SC infusion over 14 hours
  ND0612 (Levodopa/Carbidopa solution, 538/67 mg daily) + IR-LD/CD (oral Levodopa/Carbidopa, 150/15 mg in the morning)
Period: Overall Study
Arm/Group | ND0612 (Levodopa/Carbidopa Solution) Dosing Regimen 1 | ND0612 (Levodopa/Carbidopa Solution) Dosing Regimen 2
Started | 19 | 19
Completed | 16 | 17
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ND0612 Regimen 1 - 24-hr Infusion: Randomized participants received via a pump continuous, SC, 24-hour infusion of ND0612.
- ND0612 Regimen 2 - 14-hr Infusion: Randomized participants received via a pump continuous, SC, 14-hour infusion of ND0612. Infusion started at wake-up time supplemented with an oral IR LD/CD tablet.
- Total: Total of all reporting groups
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion | ND0612 Regimen 2 - 14-hr Infusion | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10.1) | 64 (8.5) | 63.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 12 | 14 | 26
Modified Hoehn and Yahr Stage [Count of Participants; unit: Participants] — A commonly used system for describing how the symptoms of Parkinson's disease progress.
  Stage 0: No signs of disease. Stage 1: Unilateral symptoms only. Stage 1.5: Unilateral and axial involvement. Stage 2: Bilateral symptoms. No impairment of balance. Stage 2.5: Mild bilateral disease with recovery on pull test. Stage 3: Balance impairment. Mild to moderate disease. Physically independent. Stage 4: Severe disability, but still able to walk or stand unassisted. Stage 5: Needing a wheelchair or bedridden unless assisted.
  Participants
    1 | 1 | 0 | 1
    1.5 | 0 | 1 | 1
    2 | 13 | 11 | 24
    2.5 | 4 | 5 | 9
    3 | 1 | 2 | 3
Time since Parkinson's disease diagnosis [Mean (Standard Deviation); unit: Years] | 10.7 (5.5) | 12.2 (5) | 11.5 (5.2)
Time since motor fluctuations [Mean (Standard Deviation); unit: Years] | 5.7 (6.9) | 5.5 (4.8) | 5.6 (5.9)
Time since dyskinesia onset [Mean (Standard Deviation); unit: years] | 3.1 (2.7) | 4.2 (3.4) | 3.7 (3.1)
Daily "OFF" time [Mean (Standard Deviation); unit: Hours] — "OFF" state is a phase with no response to medication and significant motor symptoms. An assessment of motor state ("OFF", "ON" without dyskinesia, "ON" with dyskinesia (mild, moderate, severe)) was performed by the blinded rater during 8 hours (normalized to 16 hours of awake time).
  Hours | 5.6 (2.1) | 5.0 (2.4) | 5.3 (2.2)
Daily "Good ON" time [Mean (Standard Deviation); unit: Hours] — "ON" without dyskinesia and "ON" with mild dyskinesia. An assessment of motor state ("OFF", "ON" without dyskinesia, "ON" with dyskinesia (mild, moderate, severe)) was performed by the blinded rater during 8 hours (normalized to 16 hours of awake time).
  Hours | 9.2 (3.3) | 8.5 (3.3) | 8.9 (3.2)
Daily time with troublesome dyskinesia [Mean (Standard Deviation); unit: Hours] — Dyskinesia defined as moderate or severe in intensity. An assessment of motor state ("OFF", "ON" without dyskinesia, "ON" with dyskinesia (mild, moderate, severe)) was performed by the blinded rater during 8 hours (normalized to 16 hours of awake time).
  Hours | 1.2 (2.8) | 2.5 (3.7) | 1.9 (3.3)
UPDRS Part III (motor) score [Mean (Standard Deviation); unit: Score] — Unified Parkinson's Disease Rating Scale (UPDRS) is divided into four scales. Part III (questions 18-31) is done as a motor examination. The various items to be rated are scored using a 5-point system (i.e., 0 is normal and 4 indicates a severe abnormality, half point scores are allowed for Part III questions). The range of score values is from 0 to 132. Higher value indicate greater impairment.
  Score | 37.4 (14.5) | 37.3 (13.3) | 37.3 (13.7)
PD medications [Count of Participants; unit: Participants]
  Levodopa | 19 | 19 | 38
  Dopamine agonists | 9 | 13 | 22
  Monoamine oxidase inhibitors | 11 | 10 | 21
  Amantadine | 5 | 7 | 12
  Entacapone | 2 | 4 | 6
  Trihexyphenidyl | 1 | 0 | 1
Levodopa dose [Mean (Standard Deviation); unit: mg] | 996 (552) | 948 (305) | 972 (441)

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily "OFF" Time
Description: Based on Parkinson's disease symptom assessment, "ON" time is when there is good response to medication and few symptoms. "OFF" time is when no there is no response to medication and significant motor symptoms. An "ON/OFF" Log was completed by a blinded rater starting before the first dose of LD/DDI and following the first dose at 30 min intervals for 8 hrs. The changes in "OFF" time as hours (normalized to 16 hrs of awake time) during the 8 hrs of data collection were estimated. Negative change from baseline for "OFF" time indicates improvement.
Time Frame: Baseline to Day 28
Population: mITT Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion | ND0612 Regimen 2 - 14-hr Infusion
Number analyzed (Participants) | 19 | 19
Hours | -2.8 [-4.6 to -0.9] | -1.3 [-3.1 to 0.5]

2. Secondary Outcome: The Percentage of Subjects With Full "ON" at Approximately 08:00 and Approximately 09:00, as Determined by the Subject
Description: Based on Parkinson's disease symptom assessment, "ON" time is when there is good response to medication and few symptoms. "OFF" time is when no there is no response to medication and significant motor symptoms. Subjects were asked to indicate when exactly in their opinion they had turned to full "ON" (i.e. an "ON" response comparable to the "ON" response to standard oral LD/DDI treatment). Higher percentage of subjects with full "ON" on Day 28 indicates improvement.
Time Frame: Baseline to Day 28
Population: mITT Set in Regimen 1. Regimen 2 was not optimized for morning efficacy assessment (it required the arrival of a nurse in the morning to administer oral IR LD/CD and begin the infusion).
Measure: Count of Participants; unit: Participants
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion
Number analyzed (Participants) | 19
Participants
  Baseline: Full "ON" by 8:00 | 3
  Baseline: Full "ON" by 9:00 | 7
  Day 28: Full "ON" by 8:00: number analyzed (Participants) | 16
  Day 28: Full "ON" by 8:00 | 7
  Day 28: Full "ON" by 9:00: number analyzed (Participants) | 16
  Day 28: Full "ON" by 9:00 | 13

3. Secondary Outcome: Change in Daily "Good ON" Time as Assessed by a Blinded Rater
Description: Based on Parkinson's disease symptom assessment, "ON" time is when there is good response to medication and few symptoms. "OFF" time is when no there is no response to medication and significant motor symptoms. "Good ON" time means "ON" time without troublesome dyskinesia (involuntary muscle movement), defined as the sum of "ON" time without dyskinesia and "ON" time with non-troublesome dyskinesia. An "ON/OFF" Log was completed by a blinded rater starting before the first dose of LD/DDI and following the first dose at 30 min intervals for 8 hrs. Daily total scores were normalized to 16 hours of awake time. Positive change from baseline for "ON" time without dyskinesia and for "Good ON" time, and a negative change in "ON" time with moderate or severe (troublesome) dyskinesia indicates improvement.
Time Frame: Baseline to Day 28
Population: mITT Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion | ND0612 Regimen 2 - 14-hr Infusion
Number analyzed (Participants) | 19 | 19
Hours | 3.7 [1.9 to 5.6] | 2.8 [1.0 to 4.6]

4. Secondary Outcome: Change in Morning UPDRS Part III (Motor) Scores
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. UPDRS part III (motor) score is calculated as the sum of the individual UPDRS items 18-31, each of which are measured on a 5-point scale (i.e., 0 is normal and 4 indicates a severe abnormality). UPDRS part III was done as a motor examination on Day 1 before the first dose of standard oral LD/DDI and at the same time on Day 28. The range of score values is from 0 to 132. Higher scores correlate with greater motor impairment.
Time Frame: Baseline to Day 28
Population: mITT Set
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion | ND0612 Regimen 2 - 14-hr Infusion
Number analyzed (Participants) | 19 | 19
score on a scale | -19.1 [-25.6 to -12.5] | -10.7 [-16.8 to -4.6]

5. Secondary Outcome: Change in UPDRS Part II (ADL) Scores
Description: The Unified Parkinson's disease rating scale (UPDRS) is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The UPDRS Part II (activity of daily living) score was calculated as the sum of the individual UPDRS items 5-17. The Part II score is the sum of the answers to the 13 questions that comprise Part II, each of which are measured on a 5-point scale (i.e., 0 is normal and 4 indicates a severe abnormality). The range of score values is from 0 to 52. Higher scores correlate with greater impairments for daily activities.
Time Frame: Baseline to Day 28
Population: mITT Set
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion | ND0612 Regimen 2 - 14-hr Infusion
Number analyzed (Participants) | 19 | 19
score on a scale | -2.9 [-5.4 to -0.5] | -1.9 [-4.2 to 0.4]

6. Secondary Outcome: CGI-Improvement (CGI-I) Score as Assessed by Investigator
Description: Global improvement was rated by the investigator or designee using Clinical Global Impression of Improvement (CGI-I). The CGI-I employs a 7-point scale with 1 being "very much improved" and 7 being "very much worse" for improvement rating.
Time Frame: Baseline to Day 28
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion | ND0612 Regimen 2 - 14-hr Infusion
Number analyzed (Participants) | 19 | 19
Participants
  Day 3: Subjects with improvements | 10 | 9
  Day 28: Subjects with improvements: number analyzed (Participants) | 18 | 19
  Day 28: Subjects with improvements | 14 | 13
  CGI-I score on Day 28: Very much improved: number analyzed (Participants) | 16 | 18
  CGI-I score on Day 28: Very much improved | 5 | 2
  CGI-I score on Day 28: Much improved: number analyzed (Participants) | 16 | 18
  CGI-I score on Day 28: Much improved | 6 | 7
  CGI-I score on Day 28: Minimally improved: number analyzed (Participants) | 16 | 18
  CGI-I score on Day 28: Minimally improved | 3 | 4
  CGI-I score on Day 28: No change: number analyzed (Participants) | 16 | 18
  CGI-I score on Day 28: No change | 1 | 5
  CGI-I score on Day 28: Minimally worse: number analyzed (Participants) | 16 | 18
  CGI-I score on Day 28: Minimally worse | 1 | 0
  CGI-I score on Day 28: Much worse: number analyzed (Participants) | 16 | 18
  CGI-I score on Day 28: Much worse | 0 | 0
  CGI-I score on Day 28: Very much worse: number analyzed (Participants) | 16 | 18
  CGI-I score on Day 28: Very much worse | 0 | 0

7. Secondary Outcome: Change in PDSS-2 Total Score
Description: The quality of night sleep was rated by the subjects using the Parkinson's Disease Sleep Scale (PDSS)-2, which includes questions addressing 15 commonly reported symptoms associated with sleep disturbance in PD. Each question is assessed from 0 (Always) to 10 (Never). The total score values range from 0 to 150. Higher scores indicate a lower quality of sleep, i.e., a reduction in the score indicates an improvement in sleep quality.
Time Frame: Baseline to Day 27
Population: mITT Set
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion | ND0612 Regimen 2 - 14-hr Infusion
Number analyzed (Participants) | 19 | 19
score on a scale | -4.1 [-8.0 to -0.2] | -0.8 [-4.4 to 2.9]

8. Secondary Outcome: Change in PDQ-39 Summary Index and the 8-dimension Scores
Description: Subjects were requested to rate their quality of life using the Quality of Life in Parkinson's Disease (PDQ)-39, a 39-item, self-administered questionnaire with 8 discrete dimensions (mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort.). The PDQ-39 Summary Index is the sum of the dimension scores divided by the number of dimensions. The total score values range from 0 to 100%. Higher scores indicate a worse quality of life.
Time Frame: Baseline to Day 27
Population: mITT Set
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion | ND0612 Regimen 2 - 14-hr Infusion
Number analyzed (Participants) | 19 | 19
score on a scale | -7.5 [-12.9 to -2.1] | -3.7 [-8.9 to 1.5]

9. Post Hoc Outcome: Percentage of Subjects Who Achieved at Least Certain Percent Reduction in Average Daily Normalized "OFF" Time
Description: Determination of percentage of subjects who had a complete and 50% reduction in daily "OFF" time from baseline to Day 28 during 8 hrs observations.
Time Frame: Baseline to Day 28
Population: mITT Set subjects in Regimen 1 who had valid data for the analysis at baseline and Day 28. LOCF Imputation.
Measure: Count of Participants; unit: Participants
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion
Number analyzed (Participants) | 19
Participants
  Subjects who Achieved 50% reduction in average daily normalized "OFF" time | 12
  Subjects who Achieved complete reduction in average daily normalized "OFF" | 8

ADVERSE EVENTS:
Time Frame: From Baseline to the end of treatment plus 28 days
Description: Treatment emergent adverse events are defined as all AEs that start on or after the start of first study drug administration
Arm/Group | ND0612 Regimen 1 - 24-hr Infusion | ND0612 Regimen 2 - 14-hr Infusion
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/19 | 2/19
Other Adverse Events (participants affected / at risk) | 15/19 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ND0612 Regimen 1 - 24-hr Infusion (N=19) | ND0612 Regimen 2 - 14-hr Infusion (N=19)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 — Worsening
Subcutaneous abscess (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ND0612 Regimen 1 - 24-hr Infusion (N=19) | ND0612 Regimen 2 - 14-hr Infusion (N=19)
Infusion site nodule (General disorders) | 11 | 7
Infusion site bruising (General disorders) | 4 | 3
Infusion site erythema (General disorders) | 5 | 2
Infusion site haemorrhage (General disorders) | 2 | 3
Infusion site haematoma (General disorders) | 3 | 1
Infusion site pain (General disorders) | 1 | 3
Infusion site edema (General disorders) | 1 | 1
Infusion site pruritus (General disorders) | 2 | 0
Parkinson's disease (Nervous system disorders) | 1 | 2 — Worsening
Headache (Nervous system disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.